CLINICAL TRIAL: NCT01203202
Title: A Randomized, Double-blind, Placebo-controlled, Fixed Dose, Parallel Grouped Clinical Study to Evaluate the Tolerability and to Determine the Adequate Dosage of PED-1 and PED-2 in Male Patients With Premature Ejaculation
Brief Title: Phase 2 Trial of PED-1 and PED-2 in Male Patients With Premature Ejaculation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Symyoo (Industry)
Responsible Party: Whan-Seok Choi, Seoul St. Marry's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTC PE 02
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Premature Ejaculation
Keywords: PE; IELT; DCIT
MeSH Terms: conditions — Premature Ejaculation | interventions — Clomipramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PED 0 (Placebo Comparator): placebo
  Interventions: Drug: Clomipramine
- PED 1 (Experimental): PED-1 (clomipramine 15mg)
  Interventions: Drug: Clomipramine
- PED-2 (Experimental): PED-2 (Clomipramine 30mg)
  Interventions: Drug: Clomipramine

INTERVENTIONS:
Drug: Clomipramine — 15mg and 30mg on demand
  Other Names: PED-1; PED-2

SUMMARY:
The purpose of this study is to evaluate whether PED-1 (15mg) and PED-2 (30mg) are tolerable and effective in the treatment of premature ejaculation.

DETAILED DESCRIPTION:
This study is to evaluate whether PED-1 and PED2 are tolerable and effective in the treatment of premature ejaculation. The patients will be randomized and allocated to three treatment groups into placebo, PED-1, and PED-2. The creteria for IELT for enrollment will be > or =2 min in the at least 75% of the sexual intercourse. To diagnosis premature ejaculation, the PEDT will be used. The patients ungone drug free baseline line period will take test drugs for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent for subjects and partdners
* Men 20-65
* stable monogamous relation at least for 6 mn
* PEDT more than 9
* at least 6 Mn of premature ejaculation Hx
* IELT of =< 2 min in >= 75% of evaluable events during 4 week secreening period

Exclusion Criteria:

* Hx of medical or psychiartric illness
* erectile dysfunction (<21 IIEF EF domain score) or other forms of sexual dysfunction
* Partner sexual dysfunction
* known hypersensitivity to clomipramine and contraindications for clomipramine

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Fold cahnges of Intraviginal ejaculation latency time (IELT) | 4 weeks

SECONDARY OUTCOMES:
Drug coitus interval time | 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Whan-Seok Choi, MD, PhD, Principal Investigator — Seoul St. Marry's Hospital
Locations (2):
- South Korea (2):
  - Ewha University Mok-dong Hospital, Seoul
  - Seoul St. Marry's Hospital, Seoul